CLINICAL TRIAL: NCT00247780
Title: Cavotricuspid Isthmusblock and Circumferential Pulmonary Vein Isolation in Patients With Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Heart Foundation (Other); H. Lundbeck A/S (Industry)
Responsible Party: Jacob Pontoppidan, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JAP-PV-01
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Pulmonary vein isolation; Tissue Doppler echocardiography
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Procedure: Pulmonary vein isolation and cavotricuspid ishtmusblock

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia. Pulmonary vein isolation (PVI) in the left atrium using radiofrequency energy is a new and promising non-medical treatment in patients with symptomatic AF with reported success rates of 65 % to 90 % depending on AF classification and ablation procedure. However, the risk of recurrence has led to suggestions of how to improve the clinical outcome by tailoring a more efficient ablation procedure. A prospective, randomised study with 150 patients with symptomatic AF referred for PVI has been initiated and patients are allocated to PVI alone (75 patients) or PVI with additional ablation in the right atrium (75 patients). Patients undergo extensive monitoring of the heart rhythm during follow-up to document symptomatic or asymptomatic AF or atrial flutter. The presence of asymptomatic AF after PVI could potentially affect the management of the anticoagulation therapy in these patients. The structural and functional changes in the atria after PVI is characterized by new imaging techniques (Tissue Doppler Imaging(TDI))of the atria and cardiac neurohormones. TDI may be an effective tool for characterising changes in the left atrial function after PVI. Neurohormones may provide new information regarding the changes in left atrial function and clinical outcome after PVI in patients with AF.

We hypothesize that:

* Among patients with predominant atrial fibrillation, PVI with additional ablation in the right atrium is associated with better outcome, i.e. freedom of symptomatic AF/atrial flutter overall.
* Asymptomatic AF and atrial flutter occur frequently after PVI.
* Left atrial volume and systolic function correlates to AF recurrence after PVI.
* Neurohormones levels correlates to AF recurrence after PVI.

DETAILED DESCRIPTION:
BACKGROUND:

Atrial fibrillation (AF) is the most common cardiac arrhythmia. Medical treatment is often inefficient or associated with side effects. Pulmonary vein isolation (PVI) in the left atrium using radiofrequency energy is a new and promising non-medical treatment in patients with symptomatic AF with reported success rates of 65 % to 90 % depending on AF classification and ablation procedure (1).

Circumferential PVI appears to be the superior ablation technique in patients with AF (2). However, the risk of recurrence has led to suggestions of how to improve the clinical outcome by tailoring a more efficient ablation procedure. Patients with AF often have coexisting atrial flutter (3), but it is uncertain if patients referred for PVI can benefit from additional cavotricuspid isthmusblock (CTI) which is the traditional ablation treatment of atrial flutter. A recent study indicates that PVI reduces both AF and atrial flutter by eliminating sharing triggers in the pulmonary veins (4). Other investigators showed that patients with AF and atrial flutter prior or during PVI had high risk of recurrent atrial flutter during follow-up, and that successful PVI did not reduce the risk of recurrent atrial flutter (3). The current approach in our lab is to perform additional CTI in cases of documented atrial flutter, but CTI may potentially improve the overall outcome (freedom of symptomatic arrhythmia) in patients without documented atrial flutter, especially since most symptomatic periods are undocumented.

A prospective, randomised study with 150 patients with symptomatic AF referred for PVI has been initiated and patients are allocated to PVI alone (75 patients) or PVI with additional CTI (75 patients). Patients undergo extensive Holter monitoring during follow-up to document symptomatic or asymptomatic AF or atrial flutter. Patients with AF have a high incidence of asymptomatic AF which correlates to an increased risk of tromboembolic complications (5). The presence of aymptomatic AF after PVI could potentially affect the management of the anticoagulation therapy in these patients.

The structural and functional changes in the atria after PVI have been described in few studies. To our knowledge, Tissue Doppler Imaging (TDI) and neurohormones (NT-pro-BNP and ANP) have not previously been used in characterising the left atrial function after PVI. New echocardiographic modalities such as TDI have been introduced in the characterisation of the left ventricle systolic function in ischemic heart disease and congestive heart failure. TDI has been used for characterising the global and segmental atrial systolic function in healthy individuals (6), and TDI may be an effective tool for characterising changes in the left atrial function after PVI.

Neurohormones are produced in the left ventricle/atrium, and patients with AF have elevated levels due to atrial stretch. Cardioversion from AF to sinus rhythm is associated with normalisation of the BNP/ANP levels (7), and BNP is an independent risk factor of developing AF in patients with mild congestive heart failure (8). Neurohormones may therefore provide new information regarding the changes in left atrial function and clinical outcome after PVI in patients with AF.

PURPOSE:

* To investigate the effect of additional cavotricuspid isthmusblock in patients with AF referred for circumferential pulmonary vein isolation.
* To investigate the incidence of asymptomatic AF and atrial flutter after ablation by extensive Holter monitoring.
* To characterise left atrial volume and function before and after PVI by echocardiographic assessment (TDI) and measurements of neurohormones (NT-pro-BNP and ANP).

HYPOTHESIS:

* Among patients with predominant AF, PVI with additional cavotricuspidal isthmusblock is associated with better outcome, i.e. freedom of symptomatic AF/atrial flutter overall.
* Asymptomatic AF and atrial flutter occur frequently after PVI.
* Left atrial volume and systolic function correlates to AF recurrence after PVI.
* ANP/NT-pro-BNP levels correlates to AF recurrence after PVI.

DESIGN AND MATERIALS:

A prospective, randomised study with 150 patients referred to PVI due to symptomatic paroxysmal or persistent AF. Patients are randomised to circumferential PVI with (75 patients) or without (75 patients) cavotricuspid isthmusblock in the right atrium. Follow up period of 12 months.

Eighty of the included patients (40 with paroxysmal and 40 with persistent AF) undergo TDI-echocardiography and neurohormonal measurements.

METHOD:

Admission:

* History, physical examination, medication.
* Echocardiographic characterisation of left atrial function and volume and left ventricle systolic and diastolic function (TDI in 80 patients).
* NT-pro-BNP/ANP measurements (in 80 patients).
* Questionnaire (SF-36).
* Circumferential PVI. Patients are randomised to PVI with or without cavotricuspid isthmusblock.

Ablation:

One quadripolar 5-F catheter (St. Jude Medical) is placed in the right ventricular apex and a decapolar catheter (Biosense Webster) in the coronary sinus. Transseptal access to the left atrium is achieved by the use of a SL1 sheath (St. Jude Medical). Three-dimensional maps of the left atrium are constructed with a quadripolar D-curve mapping catheter (3.5-mm Navistar, Biosense Webster) with the use of a non-fluoroscopic navigation system (CARTO, Biosense-Webster). Patients are heparinized using an initial dose of 100 IE/kg with an additional 1000 IE/hour. Radiofrequency energy is delivered via the 4-mm mapping catheter. Ablation lines are deployed circumferentially around the pulmonary veins (PV) approximately 0.5 cm from the ostia. After ablation, remapping is performed during sinus rhythm or pacing from the coronary sinus. In case of AF during ablation, patients are cardioverted to sinus rhythm before remapping. The criteria of successful ablation is the elimination of potentials > 0.1 mV within the lesions determined by voltage maps.

Ultimately, the cavotricuspid ishtmusblock is performed with the ablation catheter. The position of the catheter is established using fluoroscopy or CARTO-mapping. Ishtmusblock is verified by double potentials during coronary sinus (CS) pacing, an activation detour by pacing either side of the line, and differential pacing techniques.

Follow-up:

* 24 hours heart rhythm monitoring.
* Clinical control after 3,6 and 12 months
* 1 week Holter monitoring after 3, 6 and 12 months
* NT-pro-BNP/ANP measurements after 3 and 12 months
* Echocardiography after 3 and 12 months 2D Echocardiography M-mode of the left ventricle and atrium in parasternal view Left atrium enddiastolic and endsystolic volume using Simpson biplane in apical 4 and 2-chamber view Left ventricle enddiastolic and endsystolic volume using Simpson biplane in apical 4 and 2-chamber view Color M-mode Transmitral flow (Pulsed Wave Doppler) E- og A-peak velocity, E/A ratio og E-decelerationtime Atrial emptying fraction = A velocity time integral (VTI)/total velocity time integral (VTI)

Tissue Doppler echocardiography (TDI) Segmental atrial velocity and amplitude of right and left atrium Framerate over 100 fps

Five points in the apical 4-chamber projection:

* 2 in the right atrium (lateral annular and superior)
* 3 in the left atrium (septal annular, superior and lateral annular) Three points in the apical 2 chamber view in the left atrium (posterior annular, superior and annular anterior)

STATISTICS:

The sample size is calculated on the basis of the following assumptions:

A type 1 error and type 2 error of 5 % and 20 %, respectively, are accepted. The statistical power is 80%. Thirty-five percent of patients with AF had coexisting atrial flutter in a population who were referred to PVI (3). Patients undergoing CTI due to atrial flutter have 10 % risk of recurrence. During follow-up, 90 % versus 70 % (without CTI) of the patients are expected to be free of symptoms related to atrial flutter. Based on these parameters, the sample size is 72 patients included in each group. Overall, 150 patients are included due to expected loss of patients during follow-up.

In 2003, ninety-five patients were treated with PVI in Skejby Hospital which has increased to 150 patients in 2004. The production is expected to increase further during the following years.

PRACTICAL CONSIDERATIONS:

The PhD protocol has been approved by The Faculty of Health Science at the University of Aarhus and the Local Committee of Ethics in Aarhus. The study was initiated in December 2004 and at he moment 8 patients have been included. The Institute of Clinical Experimental Research at the University Hospital of Aarhus has donated 6 months salary to Dr. Jacob Pontoppidan.

The inclusion period is 12 months. Patients are followed 12 months. Finally, 12 months are expected for dataprocessing and publications. At least 3 publications in international peer-reviewed journals are expected.

The measurements of neurohormones are performed by the Department of Clinical Biochemistry and the biochemical laboratory at the Department of Nephrology, Skejby Hospital. The echocardiographic analyses including TDI are performed by Dr. Pontoppidan, who is experienced in this technique. The electrophysiologists in the Department of Cardiology, Skejby University Hospital of Aarhus, perform the ablation procedures as described above.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic paroxysmal or persistent atrial fibrillation where medical treatment has proven inefficient or related to sideeffects.

Exclusion Criteria:

* Prior cavotricuspid isthmus ablation (for atrial flutter) Significant valvular heart disease Congestive heart failure (NYHA class 3-4) Contraindications to antithrombic treatment with Warfarin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2004-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Symptomatic AF or atrial flutter documented by ECG or Holter monitoring from the 3rd month* after the ablation (Definition: AF > 1 minute, atrial flutter > 1 minute of typical isthmusdependent flutter).

SECONDARY OUTCOMES:
Asymptomatic AF or atrial flutter documented by ECG or Holter
Macro-reentrant left atrial flutter
Left atrial dimension
Segmental tissue velocities ad amplitude in the left and right atria
Plasma ANP/NT-pro-BNP
Quality of life-score

CONTACTS AND LOCATIONS:
Overall Officials: Peter Steen Hansen, MD, DMSc, Principal Investigator; Jens Cosedis Nielsen, MD, PhD, Principal Investigator; Steen Hvitfeldt Poulsen, MD, DMSc, Principal Investigator — Unaffilliated
Locations (1):
- Department of Cardiology, Skejby University Hospital, Aarhus, Aarhus, Denmark